CLINICAL TRIAL: NCT01268280
Title: A Phase II, Double-Blind, Randomized, Three-Way Crossover, Placebo-Controlled, Pharmacodynamic Study of CK-2017357 in Patients With Generalized Myasthenia Gravis on Standard Therapy
Brief Title: Pharmacodynamic Study of CK-2017357 in Patients With Generalized Myasthenia Gravis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed after complete treatment of 32 patients after 21 months' recruitment.
Sponsor: Cytokinetics (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 4023; 1RC3NS070670-01 (NIH)
Record Dates: First submitted 2010-12-28; First posted 2010-12-30 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — CK-2017357

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Treatment Sequence 1 (Experimental): Dosing Period 1 Placebo; Dosing Period 2 CK-2017357 250 mg; Dosing Period 3 CK-2017357 500 mg
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 2 (Experimental): Dosing Period 1 Placebo; Dosing Period 2 CK-2017357 500 mg; Dosing Period 3 CK-2017357 250 mg
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 3 (Experimental): Dosing Period 1 CK-2017357 250 mg; Dosing Period 2 Placebo; Dosing Period 3 CK-2017357 500 mg
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 4 (Experimental): Dosing Period 1 CK-2017357 250 mg; Dosing Period 2 CK-2017357 500 mg; Dosing Period 3 Placebo
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 5 (Experimental): Dosing Period 1 CK-2017357 500 mg; Dosing Period 2 Placebo; Dosing Period 3 CK-2017357 250 mg
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 6 (Experimental): Dosing Period 1 CK-2017357 500 mg; Dosing Period 2 CK-2017357 250 mg; Dosing Period 3 Placebo
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357

INTERVENTIONS:
Drug: Placebo — Matching placebo in capsules administered as a single oral dose.
Drug: 250 mg CK-2017357 — 250 mg CK-2017357 in capsules administered as a single oral dose.
  Other Names: tirasemtiv
Drug: 500 mg CK-2017357 — 500 mg CK-2017357 in capsules administered as a single oral dose.
  Other Names: tirasemitiv

SUMMARY:
The primary objective of this early-stage clinical study is to demonstrate an effect of single doses of CK-2017357 on measures of skeletal muscle function and fatigability in patients with generalized myasthenia gravis (MG).

DETAILED DESCRIPTION:
This study is a Phase II, double-blind, randomized, three-way crossover, placebo-controlled, PD study of CK-2017357 in patients with generalized MG on standard therapy. 36 to 78 patients will be randomized at approximately 15 study centers to one of six different treatment sequences. Each treatment sequence consists of three dosing periods in which patients receive single oral doses of placebo, 250 mg, and 500 mg of CK-2017357. All six treatment sequences will enroll 6 patients. A wash out period of at least 7 days (to a maximum of 10 days) will be employed between the individual doses for each patient. This study is designed to assess the effects of CK-2017357 on the standardized Quantitative Myasthenia Gravis (QMG) score, Manual Muscle Test, Myasthenia Gravis Composite Assessment (MGCA) and Forced Vital Capacity. The pharmacokinetic (PK) and pharmacodynamic (PD) relationship of CK-2017357 after two single doses will be assessed versus placebo.

ELIGIBILITY:
Inclusion criteria:

* Ability to comprehend and willing to sign an Informed Consent Form (ICF)
* Ability to understand written and oral English language
* Males and females between 18 and 80 years of age, inclusive
* Patient's signs and symptoms not better explained by another disease process
* Established diagnosis of MG defined as clinical evidence of muscle weakness and positive AChR-binding antibody titer (>0.02 nmol/L)
* Myasthenia Gravis Foundation of America (MGFA) clinical classification II or III
* Stable MG disease for 4 weeks prior to randomization
* Ability to refrain from IVIg treatments during the course of the study
* Ability to refrain from cholinesterase-inhibitors (e.g. pyridostigmine) for 12 hours before each dose
* Ability to perform all elements of the QMG
* Grade of 2 or 3 in two or more of the following muscle groups as measured by QMG: right or left arm flexion, head lift, and right or left leg raise at 45° Note: Patients may re-screen if they fail due to inadequate weakness from taking pyridostigmine within 12 hours of screening
* Body mass index (BMI) of 18.0 to 36.0 kg/m2, inclusive
* Pre-study clinical laboratory findings (including troponin I [TnI] and creatine phosphokinase [CPK]) within the normal range, or if outside of the normal range, deemed not clinically significant by the Investigator
* For female patients only: Agreement to use a double barrier during sexual intercourse (1 hormonal, plus 1 barrier method, or 2 simultaneous barrier methods) birth control (birth control pills, male condom, female condom, intrauterine device, Norplant, tubal ligation, or other sterilization procedures)
* For male patients only: Agreement either to use a condom during sexual intercourse with female partners who are of reproductive potential and to have female partners use an additional effective means of contraception (e.g., diaphragm plus spermicide, or oral contraceptives) for the duration of the study and 10 weeks after the end of the study or to abstain from sexual intercourse for the duration of the study and 10 weeks after the end of the study

Exclusion criteria:

* History of chronic degenerative, psychiatric, or neurologic disorder other than MG that can produce weakness or fatigue
* Other major chronic or debilitating illnesses within six months prior to study entry
* Hepatic insufficiency (defined as ALT or AST > 3x ULN, or total bilirubin > 3 mg/dL)
* Renal insufficiency (defined as serum creatinine > 2.5 mg/dL or receiving dialysis)
* Other myasthenic syndromes (e.g. Lambert Eaton syndrome; inherited myasthenic syndrome)
* Female patients who are premenopausal and are: (a) pregnant on the basis of a serum pregnancy test, (b) breast-feeding, or (c) not using an effective method of double barrier (1 hormonal plus 1 barrier method or 2 simultaneous barrier methods) birth control (birth control pills, male condom, female condom, intrauterine device, Norplant, tubal ligation, or other sterilization procedures)
* Receipt of IVIg or plasmapheresis treatment within 6 weeks prior to the first dose of study drug
* Changes to immunosuppressive treatments (i.e., prednisone) within 6 weeks prior to the first dose of study drug
* Rituxan treatment within 3 months prior to study entry
* Participation in any other investigational study drug or device trial in which receipt of an investigational study drug or device occurred within 30 days prior to dosing
* Any prior treatment with CK-2017357
* Recent history of alcoholism or drug abuse, or significant behavioral or psychiatric problems, or other conditions which in the Investigator's opinion may impair ability to adequately comply with the requirements of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Quantitative Myasthenia Gravis score (QMG) | 1 day
  A quantitative motor assessment of muscular weakness on a scale of 0 to 3 with 0 representing "none" and 3 representing "severe". Muscular assessments included in the overall score are effects on double vision, ptosis, facial muscles, swallowing, speech, outstretched arms and legs, forced vital capacity, hand grip strength, and ability to lift head.
Pulmonary Function Test (VC in liters) | 1 day
  Forced Vital Capacity
Manual Muscle Test (MMT) | 1 day
  Sum of strength or function values assessed by physician on the neck, shoulder, hip and ankle

SECONDARY OUTCOMES:
Characterize dose and plasma concentrations of CK-2017357 and QMG | 2 days
Characterize dose and plasma concentrations of CK-2017357 and Forced Vital Capacity (FVC) | 2 days
Characterize dose and plasma concentrations of CK-2017357 and Manual Muscle Test (MMT) | 2 days
Number of patients with adverse events | 4 weeks
Modified MG Symptom Score | 2 days
  Patients will be asked questions regarding five myasthenia gravis systems including trouble using eyes, trouble eating, difficulty speaking, trouble walking and trouble performing personal grooming needs. Each of the areas is scored 0 (none at all) to 3 (very much) and the overall score combining the score of all five areas on a scale of 0 to 15 with 0 being normal and 15 being severe weakness
Patient Global Assessment | 2 days
  Patients answer a single question as to whether they feel the same, better or worse as compared to how they felt pre-dose
Investigator Global Assessment | 2 days
  Investigator answer a single as question as to whether they think the patient appears the same, better or worse as compared to the patient's status at pre-dose

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wolff, MD, FACC, Study Director — Cytokinetics, Inc.
Locations (15):
- United States (15):
  - UCSF - Fresno, Fresno, California
  - University of California - Irvine, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - Hospital for Special Care, New Britain, Connecticut
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins, Baltimore, Maryland
  - Neurocare Center for Research, Newton, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - West Penn Allegheny Health System, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Result] Sanders DB, Rosenfeld J, Dimachkie M, Meng L, Malik FI. A Study to Evaluate Efficacy, Safety and Tolerability of Single Doses of Tirasemtiv in Patients with Myasthenia Gravis. 65th Annual Meeting of the American Academy of Neurology, San Diego, CA, March 2013